CLINICAL TRIAL: NCT00406276
Title: Phase I/II Trial of RAD001 Plus Docetaxel in Patients With Metastatic or Recurrent Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: data analysis showed insufficient drug efficacy
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Suresh S. Ramalingam, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1342-2004
Record Dates: First submitted 2006-11-17; First posted 2006-12-04 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Everolimus; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001+Docetaxel (Experimental): RAD001 in combination with Docetaxel.
  Interventions: Drug: RAD001; Drug: Docetaxel

INTERVENTIONS:
Drug: RAD001 — RAD001 will be given at a dose of 5mg/day in combination with docetaxel
Drug: Docetaxel — In combination with RAD001

SUMMARY:
This is an open-label, single-arm, Phase I/II trial to determine the safety of RAD001 in combination with docetaxel and compare the efficacy of RAD001 plus docetaxel versus published Phase II and III reports of docetaxel alone in patients with recurrent NSCLC.

DETAILED DESCRIPTION:
This is an open-label, single-arm, Phase I/II trial to determine the safety of RAD001 in combination with docetaxel and compare the efficacy of RAD001 plus docetaxel versus published Phase II and III reports of docetaxel alone in patients with recurrent NSCLC.

New agents and regimens are urgently needed for lung cancer treatment. With the development of novel agents and small molecules designed to curtail the aggressive aspects of this disease, some progress has been realized. However, much more effort and insight will be required for further real gains to be made. We propose that studying the mTOR axis, known to be abnormal in non-small cell lung cancer (NSCLC), and translating that knowledge into therapeutic adjustments can lead to meaningful advances in lung cancer treatment.

Approximately 58 patients will participate at Emory Winship Cancer Institute and Emory Crawford W. Long Hospital in Atlanta, Georgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed non-small cell lung cancer (NSCLC) which is accessible to biopsy.
* Patient must have ECOG Performance Status of 0, 1, or 2.
* Life expectancy greater than 12 weeks.
* Patient must have adequate bone marrow, renal and hepatic function as defined in the protocol.
* Completed all prior therapy at least 3 weeks prior to registration and be adequately recovered from that therapy.
* Must be at least 18 years of age.
* Meet pre-entry requirements as specified in Section 7.0.
* Female patients of child-bearing potential must have a negative serum pregnancy test prior to study entry.
* Patients of child-bearing potential must agree to use an effective form of contraception while on study and for 3 months following completion of study treatment.
* Patient must not have more than one prior chemotherapy regimen.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Exclusion Criteria:

* Chronic treatment with systemic steroids or other immunosuppressive agents.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* A known history of HIV seropositivity.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Patients with an active, bleeding diathesis or an oral anti-vitamin K medication (except low dose coumadin).
* Known hypersensitivity to everolimus, sirolimus, or any of its excipients.
* Patient is pregnant or breast-feeding.
* Patient has intercurrent illness including, but not limited to: ongoing active or severe infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, myocardial infarction within 6 months, uncontrolled diabetes mellitus, chronic liver or renal disease, active upper GI tract ulceration or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient is unable to swallow RAD001.
* History of other invasive malignancies, with the exception of non-melanoma skin cancer, if there is any evidence of the malignancy being present within the past 5 years.
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80. Symptoms may include any reaction such as bronchospasm, generalized urticaria, systolic BP ≤ 80mm Hg, and angioedema.
* Patient has received treatment with an investigational agent within 4 weeks of registration.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001+Docetaxel: Docetaxel 60 mg/m^2 given intravenously over 60 minutes on day 1 of each cycle. RAD 001 5 mg by mouth once a day on days 1-19 of each cycle.
Period: Overall Study
Arm/Group | RAD001+Docetaxel
Started | 28
Completed | 24
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | RAD001+Docetaxel
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 12
Age Continuous [Median (Full Range); unit: years] | 62 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Showing Partial Response and Stable Disease With the Combination of RAD001 and Docetaxel.
Description: Partial response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive disease (PD), taking as reference the smallest sum Longest diameter(LD) since treatment started.
Time Frame: 6 weeks
Population: 24 patients received at least 2 cycles of therapy and underwent imaging studies to assess response.
Measure: Number; unit: participants
Groups:
- Docetaxel/RAD001: Docetaxel 60 mg/m^2 given intravenously over 60 minutes on day 1 of each cycle. RAD 001 5 mg by mouth once a day on days 1-19 of each cycle.
Arm/Group | Docetaxel/RAD001
Number analyzed (Participants) | 24
participants
  Partial response | 2
  Stable disease | 15
  Disease Progression | 7

2. Primary Outcome: Time to Progression:Time Period (in Months) From Study Entry Until Disease Progression, Death, or Last Date of Contact.
Description: Period from study entry until disease progression, death, or last date of contact.
  Progressive Disease: Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 6 months
Measure: Median (Full Range); unit: Months
Arm/Group | Docetaxel/RAD001
Number analyzed (Participants) | 22
Months | 4.42 [1.1 to 6.0]

ADVERSE EVENTS:
Arm/Group | RAD001+Docetaxel
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001+Docetaxel (N=28)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
small bowel resection (Gastrointestinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
death (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001+Docetaxel (N=28)
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 4
Low albumin (Blood and lymphatic system disorders) | 3
Back pain (General disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Fatigue (Gastrointestinal disorders) | 11
Anemia (Blood and lymphatic system disorders) | 7
Cholesterol (Blood and lymphatic system disorders) | 2
Leg pain (General disorders) | 2
Alopecia (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 4
Hypertension (Cardiac disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
mucositis (Gastrointestinal disorders) | 2
Triglycerides (Blood and lymphatic system disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypocalcemia (Musculoskeletal and connective tissue disorders) | 1
Low phosphorous (Blood and lymphatic system disorders) | 2
Nail changes (Musculoskeletal and connective tissue disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 11
Low creatinine (Blood and lymphatic system disorders) | 1
thrombocytopenia (Blood and lymphatic system disorders) | 1
Weightloss (General disorders) | 1
pain (General disorders) | 3
peripheral neuropathy (Nervous system disorders) | 1
Infection (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 1
dyspnea (Blood and lymphatic system disorders) | 4
Neuropathy Sensory (Nervous system disorders) | 1
myalgia (Musculoskeletal and connective tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
elevated ALK Phosphorous (Blood and lymphatic system disorders) | 1
Low sodium (Blood and lymphatic system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
dizziness (General disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 1
headache (General disorders) | 1
neutropenia (Blood and lymphatic system disorders) | 1
Thrombosis (Blood and lymphatic system disorders) | 1
Low white blood cells count (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes